CLINICAL TRIAL: NCT04167943
Title: Indirect Pulp Capping, Direct Pulp Capping, Partial Pulpotomy, Pulpotomy of Primary Molars Using TheraCal; A Clinical Trial
Brief Title: Conservative Pulp Therapy of Primary Molars Using TheraCAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariem Wassel, Assistant professor of pediatric dentistry, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-REC R 091902
Record Dates: First submitted 2019-10-26; First posted 2019-11-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Reversible Pulpitis
Keywords: indirect pulp capping; direct pulp capping; partial pulpotomy; pulpotomy; TheraCal; primary molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- indirect pulp capping (Experimental): TheraCAL PT will be applied to affected dentin covering the pup.
  Interventions: Drug: Dual cured resin modified tricalcium silicate cement
- Direct pulp Capping (Experimental): TheraCAL PT will be applied to pinpoint pulp exposures surrounded by sound dentin.
  Interventions: Drug: Dual cured resin modified tricalcium silicate cement
- Partial Pulpotomy (Experimental): Pulp exposure will be enlarged to a depth of 1-3 mm by a sterile round diamond bur, and then TheraCAL PT will applied after hemostasis.
  Interventions: Drug: Dual cured resin modified tricalcium silicate cement
- pulpotomy (Experimental): complete removal of coronal pulp tissue will be attempted if bleeding persisted after attempting Partial pulpotomy for exposures that are not eligible for DPC. TheraCAL PT will be applied thereafter, after achieving hemostasis.
  Interventions: Drug: Dual cured resin modified tricalcium silicate cement

INTERVENTIONS:
Drug: Dual cured resin modified tricalcium silicate cement — A resin based, dual cured tricalcium silicate based cement
  Other Names: TheraCal PT

SUMMARY:
The study is a clinical trial that assesses the clinical and radiographic success rates of 3 conservative pulp therapy treatments in primary molars compared to conventional pulpotomy using a bioactive dual cured calcium silicate cement (TheraCAL PT).

DETAILED DESCRIPTION:
Participating Children will be recruited from the outpatient's clinic of pediatric dentistry department , Faculty of Dentistry Ain Shams University and will be allocated to one of the following groups; Indirect pulp capping, direct pulp capping, partial pulpotomy or pulpotomy. TheraCAL PT, a dual cured tricalcium silicate cement will be used in all groups as the pulp capping material. Children will be followed every 6 months for a period of 1 year to evaluate clinical and radiographic success.

ELIGIBILITY:
Inclusion Criteria:

* Four to six years old healthy children
* Cooperative (frankle scale + and ++)
* With at least one vital and restorable primary molar with deep caries.

Exclusion Criteria:

* History of spontaneous pain, swelling, or sinus tract
* Pathological mobility
* pain on percussion
* Furcation or periapical radiolucency
* Internal or external pathological root resorption
* Widening of periodontal membrane space
* Discontinuity of lamina dura.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in Visual and tactile clinical examination | every 6 months
  Teeth will examined for any clinical signs of irreversible pulpitis or pulp necrosis

SECONDARY OUTCOMES:
Change in Dental Periapical Radiographic examination | every 6 months
  Teeth will be examined for any radiographic signs of pulp necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Mariem Wassel, Study Director — Faculty of Dentistry, Ain Sham University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wassel M, Hamdy D, Elghazawy R. Evaluation of four vital pulp therapies for primary molars using a dual-cured tricalcium silicate (TheraCal PT): one-year results of a non-randomized clinical trial. J Clin Pediatr Dent. 2023 Mar;47(2):10-22. doi: 10.22514/jocpd.2023.004. Epub 2023 Mar 3. PMID 36890738